CLINICAL TRIAL: NCT04913922
Title: An Open-Label Phase II Study of Relatlimab (BMS-986016) With Nivolumab (BMS-936558) in Combination With 5-Azacytidine for the Treatment of Patients With Refractory/Relapsed Acute Myeloid Leukemia and Newly Diagnosed Older Acute Myeloid Leukemia Patients
Brief Title: Relatlimab With Nivolumab and 5-Azacytidine for the Treatment of AML
Acronym: AARON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Veit Bücklein, MD, Investigator, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA224-065
Record Dates: First submitted 2021-05-14; First posted 2021-06-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; relapsed; refractory; checkpoint blockade; immune checkpoint inhibition
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Azacitidine; Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination therapy (Experimental): 5-azacitidine 75 mg/m2 body surface area s.c. for 7 days nivolumab 480mg i.v. day 1 relatlimab 80-160mg i.v. day 1
  repeat day 28
  Interventions: Drug: Azacitidine Injection; Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Azacitidine Injection — s.c. 75 mg/m2 BSA for 7 days
Drug: Nivolumab — 480 mg i.v.
Drug: Relatlimab — 80-160mg i.v.

SUMMARY:
The clinical trial will test the safety and tolerability of a combination therapy (azacitidine in combination with two checkpoint inhibitors, nivolumab [Anti-PD1] and relatlimab [Anti-LAG3]) in patients with relapsed/refractory Acute Myeloid Leukemia (AML) and patients ≥ 65 years with initial diagnosis of AML.

Primary objectives are:

* maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of the combination therapy during the lead-in phase of the clinical trial (6-12 patients) and
* objective response rate (ORR) of the combination therapy in the phase II part of the study (up to 24 patients).

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (R/R AML):

- Patients with AML who have failed first line induction chemotherapy (consisting of a minimum of two intensive chemotherapy cycles, e.g. 7+3 or HAM) or patients with AML who have relapsed after achieving complete remission (CR), CRi, or CRp, or patients who have failed up to one prior salvage therapy

Cohort 2 (frontline older AML):

- Patients aged ≥65 years with previously untreated AML who are unfit for or decline standard induction therapy.

General inclusion criteria:

* Patients not eligible for intensive induction chemotherapy and/or allogeneic stem cell transplant.
* Age ≥18 years
* ECOG Performance Status ≤2
* Adequate organ function:

Total bilirubin ≤2 x ULN (≤3 × ULN if due to leukemic involvement or Gilbert's syndrome) AST and ALT ≤2.5 × ULN (≤5.0 × ULN if due to leukemic involvement) Serum creatinine ≤2 × ULN or glomerular filtration rate (GFR) ≥50 mL/h

* Adequate cardiac function: TTE with documented LVEF ≥50%
* At least 2 weeks OR at least 5 half-lives interval from prior treatment to time of initiation of study medication
* GvHD of grade ≤A on ≤10 mg prednisone without any additional immunosuppressive therapies (tacrolimus, ciclosporin, etc.)
* Written informed consent
* Negative pregnancy test and adequate methods of contraception for females of childbearing potential, adequate methods of contraception for males

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Biphenotypic or bilineage leukemia
* Known allergy or hypersensitivity to 5-azacytidine, nivolumab, relatlimab, or any of their components
* History of life-threatening toxicity related to prior immune therapy
* Previous treatment with immunotherapeutic drugs targeting PD-1/PD-L1 in combination with 5-azacytidine
* Previous treatment with LAG-3 targeted agents
* Known history of severe interstitial lung disease or severe pneumonitis
* Known history (active, known, or suspected) of any of the following autoimmune diseases:

inflammatory bowel disease rheumatoid arthritis systemic progressive sclerosis systemic lupus erythematosus autoimmune vasculitis

* Active uncontrolled pneumonitis
* Active uncontrolled infection
* Symptomatic or poorly controlled CNS leukemia
* Confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* Uncontrolled or significant cardiovascular disease
* Troponin T (TnT) or I (TnI) > 2 × institutional ULN
* Organ allografts
* Allogeneic hematopoietic stem cell transplantation within the last 100 days before first study drug administration
* Active GvHD > grade A
* Known human immunodeficiency virus seropositivity
* Known positivity for hepatitis B by surface antigen expression or active hepatitis C infection
* Other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety
* Patients unwilling or unable to comply with the protocol
* Patients who are pregnant or breastfeeding
* Prisoners and subjects who are compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | after completion of the first cycle in the fist 6-12 patients, approximately during the first 6-12 months of study conduct
  To determine the MTD of relatlimab in combination with nivolumab and 5-azacytidine in patients with R/R AML.
Dose-limiting toxicities (DLTs) | after completion of the first cycle in the fist 6-12 patients, approximately during the first 6-12 months of study conduct
  To determine the DLT of relatlimab in combination with nivolumab and 5-azacytidine in patients with R/R AML.
Objective response rate (ORR) | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To estimate the ORR to treatment with relatlimab + nivolumab + 5-azacytidine in patients with R/R AML and Patients ≥65 years with initial diagnosis of AML

SECONDARY OUTCOMES:
Hematologic improvement | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To determine the number of patients with R/R AML or Patients ≥65 years with initial diagnosis of AML treated with relatlimab + nivolumab + 5-azacytidine who have a hematologic improvement (HI) in platelets, hemoglobin, or absolute neutrophil count (ANC)
Blast reduction | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To determine the number of patients with R/R AML or Patients ≥65 years with initial diagnosis of AML treated with relatlimab + nivolumab + 5-azacytidine who have a blast reduction (defined as ≥50% reduction in blast percentage compared to baseline blast percentage in bone marrow)
Duration of response (DOR) | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To assess the duration of response (DOR) of patients with R/R AML or Patients ≥65 years with initial diagnosis of AML treated with relatlimab + nivolumab + 5-azacytidine.
Disease-free survival (DFS) | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To assess the disease-free survival (DFS) of patients with R/R AML or Patients ≥65 years with initial diagnosis of AML treated with relatlimab + nivolumab + 5-azacytidine.
Overall survival (OS) | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To assess the overall survival (OS) of patients with R/R AML or Patients ≥65 years with initial diagnosis of AML treated with relatlimab + nivolumab + 5-azacytidine.

OTHER OUTCOMES:
Immunological changes | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To study immunological changes in the peripheral blood and bone marrow in response to relatlimab + nivolumab + 5-azacytidine therapy, assessed by the frequency of T-cell (subsets), regulatory T cells, and immune checkpoint expression on blasts and T cells by flow cytometry and RNA Sequencing
Molecular changes | During Phase II expansion phase, after completion of lead-in phase, approximately during months 7-48 of study conduct
  To study the methylation status of blast DNA in the peripheral blood and bone marrow in response to relatlimab + nivolumab + 5-azacytidine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marion Subklewe, MD, Principal Investigator — Department of Medicine III, University of Munich
Locations (1):
- University Hospital, LMU Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No